CLINICAL TRIAL: NCT06777316
Title: A Phase 1/2 Study of a Selective FGFR2/3 Inhibitor, CGT4859, in Patients With Cholangiocarcinoma and Other Advanced Solid Tumors Harboring FGFR2 and/or FGFR3 Genetic Alterations
Brief Title: A Study of an FGFR2/3 Inhibitor (CGT4859) in Patients With Cholangiocarcinoma and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CGT4859-24-101
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Cholangiocarcinoma; Other Solid Tumors, Adult; FGFR2 Gene Fusion/Rearrangement; FGFR2 Gene Amplification; FGFR2 Gene Short Variants; FGFR3 Gene Fusion/Rearrangement; FGFR3 Gene Amplification; FGFR3 Gene Short Variants; FGFR2 Genetic Alterations; FGFR3 Genetic Alterations; Advanced Solid Tumors
Keywords: Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma; Advanced Solid Tumors; Investigational Drug; Phase 1; Phase 2; FGFR2; FGFR3; FGFR2/3; First in human; FGFR 2 genetic alterations; FGFR3 genetic alterations
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension

STUDY DESIGN:
Intervention Model Description: Phase 1 will evaluate multiple ascending doses until the highest safe dose and the recommended phase 2 dose (RP2D) are determined.
  Phase 2 will evaluate the RP2D in 4 cohorts defined by tumor type and prior therapy based on Phase 1 results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): Multiple doses of CGT4859 for oral administration
  Interventions: Drug: CGT4859
- Phase 2: Signal Seeking (Experimental): Oral dose of CGT4859 at the RP2D as determined in Phase 1
  Interventions: Drug: CGT4859

INTERVENTIONS:
Drug: CGT4859 — CGT4859 is a selective FGFR2/3 inhibitor

SUMMARY:
This is an open-label, phase 1/2 study evaluating the safety, tolerability, pharmacokinetic (what the body does to the drug), pharmacodynamic (what the drug does to the body), and antitumor activity of CGT4859 in adult participants with intrahepatic cholangiocarcinoma (iCCA) or other advanced solid tumors with FGFR2 and/or FGFR3 genetic alternations.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed locally advanced, metastatic, and/or unresectable iCCA or other solid tumor with documented FGFR2/3 alteration in blood and/or tumor.
2. Previously treated with, not appropriate for, or declined standard-of-care first-line treatment.
3. Have measurable disease per RECIST v1.1.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Have clinically acceptable local laboratory screening results (clinical chemistry and hematology) within certain limits.
6. Resolution of toxicities from prior therapy to ≤Grade 1 (or baseline), including resolution of clinically significant laboratory abnormalities, before the first dose of study drug. Exceptions are alopecia, hypothyroidism, or type 1 diabetes mellitus controlled with medical intervention, and paronychia controlled with local intervention.

Key Exclusion Criteria:

1. Received chemotherapy or anticancer therapies or radiotherapy within certain timeframes before first dose of study drug.
2. Major surgeries (eg, abdominal laparotomy) within 4 weeks of the first dose of study drug.
3. Clinically significant corneal or retinal disorders or current evidence of retinal detachment.
4. Received more than 2 prior FGFRi therapies
5. Active, symptomatic, or untreated brain metastases unless the participant is clinically stable and off corticosteroids for ≥2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the maximum tolerated dose (MTD) and RP2D of CGT4859 - AEs | Approximately 12 months
  Incidence, severity, and seriousness or treatment-emergent adverse events (AEs) leading to dose modification
Phase 1: Determine the maximum tolerated dose (MTD) and RP2D of CGT4859 - Laboratory results | Approximately 12 months
  Clinically significant changes or abnormalities observed from baseline in laboratory results in chemistry, hematology, and coagulation parameters
Phase 1: Determine the maximum tolerated dose (MTD) and RP2D of CGT4859 - ECG results | Approximately 12 months
  Clinically significant changes or abnormalities observed from baseline in electrocardiogram (ECG) parameters
Phase 2: Evaluate antitumor activity of CGT4859 - Objective Response Rate (ORR) | Approximately 8 months

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetics | Approximately 28 days
  Plasma concentration levels of CGT4859
Phase 1: Evaluate antitumor activity of CGT4859 - Objective Response Rate (ORR) | Approximately 8 months
Phase 1 and Phase 2: Evaluate antitumor activity of CGT4859 - Disease Control Rate (DCR) | Approximately 8 months
Phase 2: Characterize the safety of CGT4859 - AEs | Approximately 9 months
  Incidence, severity, and seriousness or treatment-emergent adverse events (AEs) leading to dose modification
Phase 2: Characterize the safety of CGT4859 - Labs, ECG | Approximately 9 months
  Changes from baseline in key laboratory results and electrocardiogram (ECG) parameters
Phase 2: Pharmacokinetics at RP2D | Approximately 28 days
  Plasma concentration levels of CGT4859

CONTACTS AND LOCATIONS:
Locations (15):
- United States (13):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Stanford Cancer Institute, Palo Alto, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Christ Hospital, Cincinnati, Ohio
  - Taussig Cancer Center - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute - University of Utah, Salt Lake City, Utah
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre - UHN, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No